CLINICAL TRIAL: NCT04197414
Title: Development of Urologic Registry for Personalized Medicine in Patients With Urological Malignancy by Analyzing Circulating Tumor DNA
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-1039
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer; Renal Cell Cancer; Bladder Cancer; Ureter Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — frozen tissue, blood, and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prostate cancer: Patients diagnosed as prostate cancer and have undergone prostatectomy
- Renal cell cancer: Patients diagnosed as renal cell cancer and have undergone partial or radical nephrectomy
- Bladder cancer: Patients diagnosed as bladder cancer and have undergone radical or partial cystectomy
- Ureter cancer: Patients diagnosed as ureter cancer and have undergone nephroureterectomy or ureterectomy

SUMMARY:
Urological malignancies such as prostate cancer and renal cell cancer in Korean population have been increased due to the aged population and the westernized lifestyles. With the advancement of sequencing technologies, use of genetic mutation profiles in cancer detection and progression has been increased. However, use of circulating tumor DNA in urological malignances have been limited and few studies have been reported. Therefore, we tried to evaluate the usefulness of circulating tumor DNA in detection and monitoring of urological malignancies in Korean population. This study aims to use circulating tumor DNA in plasma and urine for the diagnosis, disease progression monitoring and therapeutic response evaluation. This study plan includes building big databases for circulating tumor DNA of urological malignancies in Korean population and to develop optimized circulating tumor DNA platform.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed as urological malignances (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer)
* 2. Patients who have undergone surgeries due to urological malignancies in Severance Hospital, Sinchon from 2019.12 and 2029.11
* 3. Those who agree to give permission to use their human source information - 4. Those who agree with this study

Exclusion Criteria:

* 1. Those who do not agree with this study
* 2. Vulnerable participants who are likely to be vulnerable to coercion or undue influence or lack decision-making

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone surgeries with urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer) in Severance Hospital, Sinchon from 2019.12 and 2029.11 were selected.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between genetic mutations of circulating tumor DNA in plasma and urine samples and genetic mutations of primary tumor tissue samples | within 2 weeks after the surgery
  evaluate mutation profiles of circulating tumor DNA in plasma and urine samples and associate with mutation profiles of primary tumor tissue samples : evaluate the mutation frequency of specific genes in both circulating tumor DNA in plasma and urine samples in association with primary tumor tissues

SECONDARY OUTCOMES:
Correlation between circulating tumor DNA and early diagnosis and prognosis in urological malignancies | within 10 years after the surgery
  evaluate the association of circulating tumor DNA and early diagnosis of urological malignancies : evaluate the association of circulating tumor DNA and early detection of recurrence : evaluate the association of circulating tumor DNA and cancer-specific survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Urological Science Institute, Yonsei University, Colleage of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No